CLINICAL TRIAL: NCT03444285
Title: Analysis on the Effects of Two Types of Warm up in Athletes With a Previous Hamstring Injury
Brief Title: Effects of Warm up in Athletes With Previous Hamstring Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Extremadura (Other)
Collaborators: Luis Espejo Antúnez (Unknown)
Responsible Party: Principal Investigator, Javier Gutiérrez Coronado, Principal Investigator, University of Extremadura
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19731973
Record Dates: First submitted 2018-02-02; First posted 2018-02-23 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Previous Hamstring Injury
Keywords: Thermotherapy; warm-up; extensibility; pain; athletes
MeSH Terms: conditions — Hyperthermia; Pain | interventions — Warm-Up Exercise

STUDY DESIGN:
Intervention Model Description: Two groups. One realize an static warm-up and the other a dynamic warm-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warm Up (Active Comparator)
  Interventions: Other: Warm Up
- Hot Pack (Active Comparator)
  Interventions: Other: Hot Pack

INTERVENTIONS:
Other: Warm Up — Run on a treadmill during 10 minutes without fatigue of the participant after this time.
  Arms: Warm Up
Other: Hot Pack — 20 minutes of hot-pack on both hamstring
  Arms: Hot Pack

SUMMARY:
The objectives of this study is to determine the immediate and 10 minutes follow-up effects of a warm-up based on a continous run on a treadmill or the application of a hot-pack in athletes with previous hamstring injury. The investigators have as an hypothesis that the subjects, after one of this interventions show statistically significant improvements in the measurements of pain, flexibility, proprioception and postural control

ELIGIBILITY:
Inclusion Criteria:

* To be 18-27 years old
* To do sports as a minimum of 5 hours per week.
* To have done sport in the last 2 years
* Have a hamstring flexibility of ≤80º on Kendall test
* Diagnosed hamstring injury the last year

Exclusion Criteria:

* To take drugs that alter the motor o postural control
* To do a program of stretching of the hamstring
* To have lumbar pain
* Recent abdominal or spinal surgery intervention

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2017-12-04 (Actual); Study Completion 2019-07-23 (Actual)

PRIMARY OUTCOMES:
Range of movement | Changes from baseline at immediately after and at 10 minutes after the intervention
  degrees
Pain | Changes from baseline at immediately after and at 10 minutes after the intervention
  Visual Analogue Scale. From 0 (not pain) to 10 (maximum pain in the world)

SECONDARY OUTCOMES:
Pressure pain threshold (PPT) | Changes from baseline at immediately after and at 10 minutes after the intervention
  Measurement of the pressure (kg/cm2) with an algometer
Joint Position Sense | Changes from baseline at immediately after and at 10 minutes after the intervention
  Degrees

CONTACTS AND LOCATIONS:
Overall Officials: Javier Gutiérrez Coronado, Physioterapist, Study Director
Locations (1):
- Universidad de Extremadura, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: No